CLINICAL TRIAL: NCT04567550
Title: A Phase 2, Randomized, Controlled, Dose-escalation Study to Evaluate the Efficacy, Safety, and Tolerability of RGX-314 Gene Therapy Delivered Via a Single Suprachoroidal Space (SCS) Injections in Participants With Diabetic Retinopathy (DR) With and Without Center Involved-Diabetic Macular Edema (CI-DME)(ALTITUDE)
Brief Title: RGX-314 Gene Therapy Administered in the Suprachoroidal Space for Participants With Diabetic Retinopathy (DR) With and Without Center Involved-Diabetic Macular Edema (CI-DME)
Acronym: ALTITUDE®
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGX-314-2202 (M23-414)
Record Dates: First submitted 2020-09-15; First posted 2020-09-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Retinopathy (DR); Center-Involved Diabetic Macular Edema (CI-DME)
Keywords: DR; CI-DME
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Steroids; aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Part 1: Observation Control Arm (No Intervention): Observation Control
- Part 1: ABBV-RGX-314 Treatment Arm (Dose 1) (Experimental): ABBV-RGX-314 Dose 1
  Interventions: Genetic: ABBV-RGX-314 Dose 1
- Part 1: ABBV-RGX-314 Treatment Arm (Dose 2) (Experimental): ABBV-RGX-314 Dose 2
  Interventions: Genetic: ABBV-RGX-314 Dose 2
- Part 1: ABBV-RGX-314 Treatment Arm (Dose 3) and Topical Steroid (Experimental): ABBV-RGX-314 Dose 3 and Topical Steroid
  Interventions: Genetic: ABBV-RGX-314 Dose 3; Drug: Topical Steroid
- Part 2: ABBV-RGX-314 Treatment Arm (Dose 4) and Topical Steroid (Experimental): ABBV-RGX-314 Dose 4 and Topical Steroid
  Interventions: Drug: Topical Steroid; Genetic: ABBV-RGX-314 Dose 4
- Part 2: Aflibercept Control (Active Comparator): Control treatment arm
  Interventions: Biological: Aflibercept

INTERVENTIONS:
Genetic: ABBV-RGX-314 Dose 1 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 1)
  Other Names: Genetic/ Combination Product
  Arms: Part 1: ABBV-RGX-314 Treatment Arm (Dose 1)
Genetic: ABBV-RGX-314 Dose 2 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 2)
  Other Names: Genetic/ Combination Product
  Arms: Part 1: ABBV-RGX-314 Treatment Arm (Dose 2)
Genetic: ABBV-RGX-314 Dose 3 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 3)
  Other Names: Genetic/ Combination Product
  Arms: Part 1: ABBV-RGX-314 Treatment Arm (Dose 3) and Topical Steroid
Drug: Topical Steroid — Topical Steroid
  Arms: Part 1: ABBV-RGX-314 Treatment Arm (Dose 3) and Topical Steroid; Part 2: ABBV-RGX-314 Treatment Arm (Dose 4) and Topical Steroid
Genetic: ABBV-RGX-314 Dose 4 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 4)
  Other Names: Genetic/ Combination Product
  Arms: Part 2: ABBV-RGX-314 Treatment Arm (Dose 4) and Topical Steroid
Biological: Aflibercept — Aflibercept
  Arms: Part 2: Aflibercept Control

SUMMARY:
ABBV-RGX-314 is being developed as a novel, potential one-time gene therapy treatment for the treatment of Diabetic Retinopathy (DR) with and without Center-Involved Diabetic Macular Edema (CI-DME). DR is a chronic and progressive complication of diabetes mellitus. It is a sight-threatening disease characterized in the early stages by neuronal and vascular dysfunction in the retina, and later by neovascularization that leads to further deterioration of functional vision. Despite the availability of current treatments, diabetic retinopathy remains the leading cause of vision loss in working-age adults, those between the ages of 20 and 74. Existing treatment with anti-VEGF agents, although shown to be effective, are limited by short therapeutic half-lives, which then require frequent intravitreal injections over the patient's lifetime, resulting in increased risk of associated adverse events and significant treatment burden. Due to the burden of treatment, patients often do not closely adhere to treatment regimens and experience sub-optimal outcomes and a decline in vision.

DETAILED DESCRIPTION:
This phase 2, randomized, dose-escalation study is designed to evaluate the efficacy, safety and tolerability of ABBV-RGX-314 gene therapy in subjects with DR with and without center-involved diabetic macular edema (CI-DME).

Part 1: For subjects with DR without CI-DME, approximately 100 participants who meet the inclusion/exclusion criteria will be enrolled into one of 5 cohorts. Participants will be randomized in Cohorts 1, 2, 4 and 5 to receive ABBV-RGX-314 or to be observed, and participants enrolled in Cohort 3 will receive ABBV-RGX-314. Cohort 1 will evaluate ABBV-RGX-314 Dose 1, Cohorts 2 and 3 will evaluate ABBV-RGX-314 Dose 2, and Cohorts 4 and 5 will evaluate ABBV-RGX-314 Dose 3. Following SCS ABBV-RGX-314 administration, participants in Cohorts 4 and 5 will receive a protocol-mandated post-procedure steroid regimen for 7 weeks. Participants who are randomized to be observed in Cohorts 1, 2, 4 and 5 will be offered ABBV-RGX-314 after completing the study.

Part 2: For subjects with DR with CI-DME, approximately 30 participants who meet the inclusion/exclusion criteria will be enrolled into one cohort (Cohort A). Participants will be randomized to receive ABBV-RGX-314 or Aflibercept Control. Cohort A will evaluate ABBV-RGX-314 Dose 4. Participants randomized to receive SCS ABBV-RGX-314 will receive a protocol-mandated course of steroid. Participants who are randomized to the Aflibercept Control arm will be offered ABBV-RGX-314 after completing the study.

ELIGIBILITY:
Part 1 (DR without CI-DME):

Inclusion Criteria:

* Patients 25-89 years of age with a diabetic retinopathy (DR) diagnosis of nonproliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy (PDR) secondary to diabetes mellitus Type 1 or 2 for which PRP or anti-VEGF injections can be safely deferred for at least 6 months
* HbA1c < 12%.
* Best corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in the study eye of ≥69 letters (approximate Snellen equivalent of 20/40 or better).
* Prior history of CI-DME in the study eye is acceptable.
* Must be willing and able to provide written, signed informed consent.

Exclusion Criteria:

* Neovascularization in the study eye from a cause other than DR.
* Presence of any active CI-DME.
* Active or history of retinal detachment in the study eye.
* Any evidence or documented history of PRP or retinal laser in the study eye.
* Patients who had a prior vitrectomy surgery.
* Women of childbearing potential.

Part 2 (DR with CI-DME):

Inclusion Criteria:

* Patients 25-89 years of age with diabetic retinopathy secondary to diabetes mellitus Type 1 or 2.
* HbA1c < 12%
* Macular thickening secondary to DME involving the center of the fovea, CST on SD-OCT (≥ 325 μm)
* Best corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in the study eye of 78-25 letters (approximate Snellen equivalent of 20/32 to 20/320)
* Participants must have demonstrated a meaningful response to anti-VEGF therapy.
* Must be willing and able to provide written, signed informed consent

Exclusion Criteria:

* Neovascularization in the study eye from a cause other than DR.
* Active or history of retinal detachment in the study eye.
* Any evidence or documented history of PRP or retinal laser in the study eye.
* Patients who had a prior vitrectomy surgery.
* Women of childbearing potential.

Note: Other inclusions/exclusions criteria apply.

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: Proportion of participants achieving a 2-step or greater improvement in DR in the study eye per the ETDRS-DRSS on 4 widefield digital stereoscopic fundus photography at Week 48 | At Week 48
  To evaluate the effect of ABBV-RGX-314 on DR by the ETDRS DRSS at Week 48.
Part 2: Mean change from baseline in Best Corrected Visual Acuity (BCVA) in the study eye at Week 54. | At Week 54
  To evaluate the effect of ABBV-RGX-314 on BCVA at Week 54.

SECONDARY OUTCOMES:
Part 1: Proportion of participants achieving an improvement in DR in the study eye per the ETDRS DRSS on 4 widefield digital stereoscopic fundus photography. | At Week 4, Week 12, Week 24, and Week 36
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1:Proportion of participants achieving a 0-step (no change) or greater improvement in DR in the study eye per the ETDRS DRSS on 4 widefield digital stereoscopic fundus photography. | At Week 4, Week 12, Week 24, Week 36, and Week 48
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1:Proportion of participants with a worsening in DR in the study eye per the ETDRS-DRSS on 4 widefield digital stereoscopic fundus photography. | At Week 4, Week 12, Week 24, Week 36, and Week 48
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1: Proportion of participants in the NPDR and PDR subgroups at baseline achieving an improvement or worsening in DR in the study eye per the ETDRS-DRSS on 4 widefield digital stereoscopic fundus photography. | At Week 4, Week 12, Week 24, Week 36, and Week 48
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1: Proportion of participants graded as proliferative diabetic retinopathy (PDR) in the study eye at baseline achieving regression to nonproliferative diabetic retinopathy (NPDR) in the study eye. | At Week 24, Week 36, and Week 48
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1: Proportion of participants achieving a 0-step (no change) or greater improvement in DR in the study eye per the ETDRS-DRSS on 4-widefield digital stereoscopic fundus photography | At Week 54, Week 62, and Week 74 (Crossover (CO) participants)
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1: Proportion of participants with a worsening in DR in the study eye per the ETDRS-DRSS on 4 widefield digital stereoscopic fundus photography. | At Week 54, Week 62, and Week 74 (Crossover participants)
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1: Mean change from baseline in the study eye in ETDRS-DRSS severity steps at Week 12, Week 24, Week 36, and Week 48 and (CO participants) change from Week 48 at Week 54, Week 62, and Week 74 | Baseline to Week 12, Week 24, Week 36, and Week 48; Week 48 to Week 54, Week 62, and Week 74 (Crossover participants)
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time.
Part 1: Incidences of overall and ocular AEs | Through Week 48; and through Week 74 (Crossover participants)
  To assess the safety and tolerability of ABBV-RGX-314
Part 1: Vector shedding analysis in serum, urine, and tears | Through Week 48; and through Week 74 (Crossover participants)
  To assess the safety and tolerability of ABBV-RGX-314
Part 1: Proportion of participants who experience ocular inflammation in the study eye following Suprachoroidal Space (SCS) ABBV-RGX-314 administration. | Through Week 48; and through Week 74 (Crossover participants)
  To evaluate the incidences of ocular inflammation following SCS ABBV-RGX-314 administration.
Part 1: Proportion of participants requiring any additional intervention in the study eye for ocular diabetic complications | Through Week 48 or Week 74 (Crossover participants)
  To evaluate the need for additional Standard of Care (SOC) intervention due to ocular diabetic complications
Part 1: Proportion of participants with any sight threatening ocular diabetic complications in the study eye based on duration of time to development of sight threatening ocular conditions | Day 1 to Week 48; Week 50 to Week 74 (Crossover participants)
  To evaluate the need for additional Standard of Care (SOC) intervention due to ocular diabetic complications
Part 1:Proportion of participants developing ocular diabetic complications in the study eye requiring treatment per SOC based on number of treatments received and duration of time from intervention to first treatment per SOC | Day 1 to Week 48; Week 50 to Week 74 (Crossover participants)
  To evaluate the need for additional Standard of Care (SOC) intervention due to ocular diabetic complications
Part 1: Proportion of participants developing ocular diabetic complications in the study eye requiring treatment per SOC based on duration of time from study intervention to first treatment and proportion of participants requiring more than 1 treatment | Day 1 to Week 48; or Week 50 to Week 74 (Crossover participants)
  To evaluate the need for additional Standard of Care (SOC) intervention due to ocular diabetic complications
Part 1: Proportion of participants developing ocular diabetic complications in the study eye requiring surgical intervention per SOC based on duration of time from study intervention to surgical intervention | Day 1 to Week 48; or Week 50 to Week 74 (Crossover participants)
  To evaluate the need for additional Standard of Care (SOC) intervention due to ocular diabetic complications
Part 1: Aqueous ABBV-RGX-314 TP concentration at assessed time points | Through Week 48 or Week 74 (Crossover participants)
  To measure aqueous ABBV-RGX-314 TP concentrations
Part 1: Serum ABBV-RGX-314 TP concentration at assessed time points | Through Week 48 or Week 74 (Crossover participants)
  To measure serum ABBV-RGX-314 TP concentrations
Part 2: Mean change from baseline in BCVA in the study eye over time | Through Week 54
  To evaluate the effect of ABBV-RGX-314 on BCVA over time
Part 2: Proportion of participants with improved BCVA in the study eye over time | Through Week 54
  To evaluate the effect of ABBV-RGX-314 on BCVA over time
Part 2: Proportion of participants with a worsening in DR in the study eye per the ETDRS-DRSS on 4 widefield digital stereoscopic fundus photography | At Week 14, Week 30, Week 38, and Week 54
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time
Part 2: Proportion of participants achieving an improvement in DR in the study eye per the ETDRS-DRSS on 4 widefield digital stereoscopic fundus photography | At Week 14, Week 30, Week 38, and Week 54
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time
Part 2: Proportion of participants achieving a 0-step (no change) or greater improvement in DR in the study eye per the ETDRS-DRSS on 4 widefield digital stereoscopic fundus photography | At Week 66 and Week 82 (Crossover participants)
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time
Part 2: Proportion of participants with a worsening in DR in the study eye per the ETDRS-DRSS on 4-widefield digital stereoscopic fundus photography | At Week 66 and Week 82 (Crossover participants)
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time
Part 2: Mean change from baseline in the study eye in ETDRS-DRSS severity steps at Week 22, Week 38, and Week 54 and (CO participants) change from Week 56 at Week 74 and Week 82 | Baseline to Week 22, Week 38, and Week 54; Week 56 to Week 74 and Week 82 (Crossover participants)
  To evaluate the effect of ABBV-RGX-314 on DR (ETDRS-DRSS) over time
Part 2: Proportion of participants with an absence of CI-DME in the study eye | At Week 54
  To evaluate the effect of ABBV-RGX-314 on CST (as determined by SD-OCT measurement) at Week 54.
Part 2: Incidences of overall and ocular AEs | Through Week 54 or Week 82 (Crossover participants)
  To assess the safety and tolerability of ABBV-RGX-314
Part 2: Vector shedding analysis in serum, urine, and tears | Through Week 54 or Week 82 (Crossover participants)
  To assess the safety and tolerability of ABBV-RGX-314
Part 2: Proportion of participants who experience ocular inflammation in the study eye following SCS ABBV-RGX-314 administration | Through Week 54 or Week 82 (Crossover participants)
  To evaluate the incidences of ocular inflammation following SCS ABBV-RGX-314 administration
Part 2: Proportion of participants requiring any additional intervention in the study eye for ocular diabetic complications to Week 54 and (CO participants) Week 82 | Through Week 54 or Week 82 (Crossover participants)
  To evaluate the need for additional SOC intervention due to ocular diabetic complications
Part 2: Proportion of participants with any sight threatening ocular diabetic complications in the study eye based on duration of time to development of sight-threatening ocular conditions | Day 1 to Week 54; Week 56 to Week 82 (Crossover participants)
  To evaluate the need for additional SOC intervention due to ocular diabetic complications
Part 2: Proportion of participants developing ocular diabetic complications in the study eye requiring treatment per SOC based on number of treatments received and duration of time from study intervention to first treatment per SOC | Day 1 to Week 54; Week 56 to Week 82 (Crossover participants)
  To evaluate the need for additional SOC intervention due to ocular diabetic complications
Part 2: Proportion of participants developing ocular diabetic complications in the study eye requiring treatment per SOC based on duration of time from study intervention to first treatment and proportion of participants requiring more than 1 treatment | Day 1 to Week 54; Week 56 to Week 82 (Crossover participants)
  To evaluate the need for additional SOC intervention due to ocular diabetic complications
Part 2: Proportion of participants developing ocular diabetic complications in the study eye requiring surgical intervention per SOC | Day 1 to Week 54; Week 56 to Week 82 (Crossover participants)
  To evaluate the need for additional SOC intervention due to ocular diabetic complications
Part 2: Mean change from baseline in CST in the study eye on SD OCT at Week 30 and Week 54 | At Week 30 and Week 54
  To evaluate the effect of ABBV-RGX-314 on anatomic outcomes assessed using SD-OCT in all ABBV-RGX-314 treated participants
Part 2: Mean change from Week 54 in CST in the study eye on SD OCT at Week 82 (Crossover participants) | At Week 82
  To evaluate the effect of ABBV-RGX-314 on anatomic outcomes assessed using SD-OCT in all ABBV-RGX-314 treated participants
Part 2: Proportion of participants achieving a reduction in CST in the study eye on SD-OCT at Week 30 and Week 54 | At Week 30 and Week 54
  To evaluate the effect of ABBV-RGX-314 on anatomic outcomes assessed using SD-OCT in all ABBV-RGX-314 treated participants
Part 2: Aqueous ABBV-RGX-314 TP concentration at assessed time points | Through Week 54 or Week 82 (Crossover participants)
  To measure aqueous ABBV-RGX-314 TP concentrations
Part 2: Serum ABBV-RGX-314 TP concentration at assessed time points | Through Week 54 or Week 82 (Crossover participants)
  To measure serum ABBV-RGX-314 TP concentrations

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - California Eye Specialists Medical Group, Inc, Pasadena, California
  - Retinal Consultants San Diego, Poway, California
  - California Retina Consultants, Santa Barbara, California
  - Southeast Retina Center, PC, Augusta, Georgia
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Wilmer Eye Institute/Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - NJ Retina, Teaneck, New Jersey
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Duke University Eye Center, Durham, North Carolina
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Charles Retina Institute, P.C., Germantown, Tennessee
  - Retina Research Institute of Texas, LLC, Abilene, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Star Retina, Burleson, Texas
  - Retinal Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No